CLINICAL TRIAL: NCT04285476
Title: Study of the Predictive Value of a Signature of microRNA in Thyroid Cytologies of Undetermined Type
Brief Title: Predictive Value of microRNA in Thyroid Cytologies of Undetermined Type
Acronym: PREDICYTHY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROCIM 2020-02 PRE
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Signature of microRNA (Experimental): Signature of miRNA in patients with Thyroid Cytologies of undetermined type and with a Bethesda classification 3, 4 or 5
  Interventions: Diagnostic Test: Signature of microRNA for patients with bethesda classification 3, 4 or 5

INTERVENTIONS:
Diagnostic Test: Signature of microRNA for patients with bethesda classification 3, 4 or 5 — If the cytology results are Bethesda 3, 4 or 5, then a miRNA analysis will be performed.

SUMMARY:
The aim is to validate a signature of microRNA (micro Ribonucleic acid) based in a first exploratory study allowing the stratification of the cytologies of indeterminate type and to study and select others. In a first step, the teams will focus on standardising the pre-analytical stages and defining a threshold of positivity. The results of microRNA signature on a cohort of 70 patients will be compared with the ultrasound and then histological data of the resection specimen.

DETAILED DESCRIPTION:
Morphological analysis of fine-needle aspiration cytology (FNAC) under ultrasound classifies thyroid nodules in 6 categories (Bethesda classification). The diagnostic approach is codified by the Society of Endocrinology and for cytologies of indeterminate type (Bethesda 3, 4 and 5), surgery of thyroid nodules is currently recommended. However, only 15.9% of the cytologies classified Bethesda 3, 26.1% of the Bethesda IV and 75.2% of the Bethesda V are actually cancers in the definitive histological analysis on surgical resection.

Thus, new tools for predicting the risk of thyroid nodule malignancy need to be developed.

To date, various risk stratification biomarkers have been reported in the literature but have not been validated in independent cohorts, thus excluding their implementation in daily practice.

In addition, two commercial nucleic acid tests are proposed at a cost not compatible with generalized diffusion. The first approach is based on a next generation sequencing analysis of a target gene panel at the nucleotide sequence or transcribed level. The second alternative combines an analysis at level 1) of the deoxyribonucleic acid (DNA) with the search for somatic variations such as mutations in oncogenes or the presence of fusion genes, and 2) microRNA with the measurement of their level of expression.

Due to their stability, their ability to modulate the expression of various messenger RNA, microRNA are an attractive line of research.

The aim is to validate a signature of microRNA based in a first exploratory study allowing the stratification of the cytologies of indeterminate type and to study and select others. In a first step, the teams will focus on standardising the pre-analytical stages and defining a threshold of positivity. The results of microRNA signature on a cohort of 70 patients will be compared with the ultrasound and then histological data of the resection specimen.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman whose Age is ≥ 18 years
2. Patient requiring ultrasound for thyroid nodule scanning with established indication of FNAC
3. Patient with Bethesda 3, 4 and 5 thyroid nodule
4. Informed patient and signed informed consent received
5. Patient affiliated to a French medical coverage system

Exclusion Criteria:

1. Patient under guardianship, curatorship or safeguarding of justice
2. Patient whose medical or psychological conditions do not permit them to complete the study or to sign the consent,
3. Patient with metastatic cancer distinct from thyroid cancer
4. Patient who has stopped treatment (chemotherapy / immunotherapy) for cancer for less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Area under receiver operating characteristic (ROC) curve of the microRNA signature | 24 months

SECONDARY OUTCOMES:
Sensitivity of the test (microRNA) | 24 months
  Sensitivity is defined as the proportion of patients with a malignant nodule (diagnosed by the gold standard method) and a positive test with miRNA signature.
Specificity of the test (microRNA) | 24 months
  The specificity of the test is defined as the proportion of patients with a benign nodule (diagnosed by the gold standard method) and a negative test with miRNA signature.
Positive predictive value (PPV) of the test (microRNA) | 24 months
  The positive predictive value is defined as the probability that the patient with a positive test is actually affected by a malignant nodule (diagnosed by the gold standard method).
Negative predictive value (NPV) of the test (microRNA) | 24 months
  The negative predictive value is defined as the probability that the patient with a negative test is actually affected by a benign nodule (diagnosed by the gold standard method).

CONTACTS AND LOCATIONS:
Overall Officials: Thierry GALVEZ, MD, Study Chair — Institut régional du Cancer de Montpellier
Locations (3):
- France (3):
  - CHU de Toulouse, Toulouse, Haute-Garonne
  - Institut régional du Cancer de Montpellier, Montpellier, Hérault
  - CHU de Nîmes, Nîmes

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients All participant data collected during the trial, after encoding with an inclusion number, 1st letter of the name and surname may be shared.
  The data of the participants will be available upon request and with the completion of a contract between the promoter and the applicant.
  The study protocol, the statistical analysis plan (PAS) and the analytical code may also be subject to data sharing as part of a transfer contract (RGPD)

REFERENCES:
- [Background] Jacques C, Guillotin D, Fontaine JF, Franc B, Mirebeau-Prunier D, Fleury A, Malthiery Y, Savagner F. DNA microarray and miRNA analyses reinforce the classification of follicular thyroid tumors. J Clin Endocrinol Metab. 2013 May;98(5):E981-9. doi: 10.1210/jc.2012-4006. Epub 2013 Apr 8. PMID 23569218
- [Background] Russ G, Bonnema SJ, Erdogan MF, Durante C, Ngu R, Leenhardt L. European Thyroid Association Guidelines for Ultrasound Malignancy Risk Stratification of Thyroid Nodules in Adults: The EU-TIRADS. Eur Thyroid J. 2017 Sep;6(5):225-237. doi: 10.1159/000478927. Epub 2017 Aug 8. PMID 29167761
- [Background] Paschke R, Cantara S, Crescenzi A, Jarzab B, Musholt TJ, Sobrinho Simoes M. European Thyroid Association Guidelines regarding Thyroid Nodule Molecular Fine-Needle Aspiration Cytology Diagnostics. Eur Thyroid J. 2017 Jul;6(3):115-129. doi: 10.1159/000468519. Epub 2017 May 19. PMID 28785538
- [Background] Cantara S, Marzocchi C, Pilli T, Cardinale S, Forleo R, Castagna MG, Pacini F. Molecular Signature of Indeterminate Thyroid Lesions: Current Methods to Improve Fine Needle Aspiration Cytology (FNAC) Diagnosis. Int J Mol Sci. 2017 Apr 6;18(4):775. doi: 10.3390/ijms18040775. PMID 28383480
- [Background] Sahli ZT, Smith PW, Umbricht CB, Zeiger MA. Preoperative Molecular Markers in Thyroid Nodules. Front Endocrinol (Lausanne). 2018 Apr 18;9:179. doi: 10.3389/fendo.2018.00179. eCollection 2018. PMID 29720964
- [Background] Dedhia PH, Rubio GA, Cohen MS, Miller BS, Gauger PG, Hughes DT. Potential effects of molecular testing of indeterminate thyroid nodule fine needle aspiration biopsy on thyroidectomy volume. World J Surg. 2014 Mar;38(3):634-8. doi: 10.1007/s00268-013-2430-x. PMID 24435929
- [Background] Nikiforov YE, Seethala RR, Tallini G, Baloch ZW, Basolo F, Thompson LD, Barletta JA, Wenig BM, Al Ghuzlan A, Kakudo K, Giordano TJ, Alves VA, Khanafshar E, Asa SL, El-Naggar AK, Gooding WE, Hodak SP, Lloyd RV, Maytal G, Mete O, Nikiforova MN, Nose V, Papotti M, Poller DN, Sadow PM, Tischler AS, Tuttle RM, Wall KB, LiVolsi VA, Randolph GW, Ghossein RA. Nomenclature Revision for Encapsulated Follicular Variant of Papillary Thyroid Carcinoma: A Paradigm Shift to Reduce Overtreatment of Indolent Tumors. JAMA Oncol. 2016 Aug 1;2(8):1023-9. doi: 10.1001/jamaoncol.2016.0386. PMID 27078145
- [Background] Faquin WC, Wong LQ, Afrogheh AH, Ali SZ, Bishop JA, Bongiovanni M, Pusztaszeri MP, VandenBussche CJ, Gourmaud J, Vaickus LJ, Baloch ZW. Impact of reclassifying noninvasive follicular variant of papillary thyroid carcinoma on the risk of malignancy in The Bethesda System for Reporting Thyroid Cytopathology. Cancer Cytopathol. 2016 Mar;124(3):181-7. doi: 10.1002/cncy.21631. Epub 2015 Oct 12. PMID 26457584
- [Background] Paulson VA, Shivdasani P, Angell TE, Cibas ES, Krane JF, Lindeman NI, Alexander EK, Barletta JA. Noninvasive Follicular Thyroid Neoplasm with Papillary-Like Nuclear Features Accounts for More Than Half of "Carcinomas" Harboring RAS Mutations. Thyroid. 2017 Apr;27(4):506-511. doi: 10.1089/thy.2016.0583. Epub 2017 Feb 24. PMID 28114855
- [Background] Strickland KC, Howitt BE, Marqusee E, Alexander EK, Cibas ES, Krane JF, Barletta JA. The Impact of Noninvasive Follicular Variant of Papillary Thyroid Carcinoma on Rates of Malignancy for Fine-Needle Aspiration Diagnostic Categories. Thyroid. 2015 Sep;25(9):987-92. doi: 10.1089/thy.2014.0612. Epub 2015 Jul 29. PMID 26114752
- [Background] Nabhan F, Porter K, Lupo MA, Randolph GW, Patel KN, Kloos RT. Heterogeneity in Positive Predictive Value of RAS Mutations in Cytologically Indeterminate Thyroid Nodules. Thyroid. 2018 Jun;28(6):729-738. doi: 10.1089/thy.2017.0635. Epub 2018 May 16. PMID 29665745
- [Background] Finoux AL, Chartrand P. [Oncogenic and tumour suppressor microRNAs]. Med Sci (Paris). 2008 Dec;24(12):1049-54. doi: 10.1051/medsci/200824121049. French. PMID 19116113
- [Background] Boufraqech M, Klubo-Gwiezdzinska J, Kebebew E. MicroRNAs in the thyroid. Best Pract Res Clin Endocrinol Metab. 2016 Oct;30(5):603-619. doi: 10.1016/j.beem.2016.10.001. Epub 2016 Nov 1. PMID 27923454
- [Background] Dom G, Frank S, Floor S, Kehagias P, Libert F, Hoang C, Andry G, Spinette A, Craciun L, de Saint Aubin N, Tresallet C, Tissier F, Savagner F, Majjaj S, Gutierrez-Roelens I, Marbaix E, Dumont JE, Maenhaut C. Thyroid follicular adenomas and carcinomas: molecular profiling provides evidence for a continuous evolution. Oncotarget. 2017 Dec 8;9(12):10343-10359. doi: 10.18632/oncotarget.23130. eCollection 2018 Feb 13. PMID 29535811
- [Background] Titov SE, Demenkov PS, Ivanov MK, Malakhina ES, Poloz TL, Tsivlikova EV, Ganzha MS, Shevchenko SP, Gulyaeva LF, Kolesnikov NN. Selection and validation of miRNAs as normalizers for profiling expression of microRNAs isolated from thyroid fine needle aspiration smears. Oncol Rep. 2016 Nov;36(5):2501-2510. doi: 10.3892/or.2016.5113. Epub 2016 Sep 20. PMID 27666315
- [Background] Lithwick-Yanai G, Dromi N, Shtabsky A, Morgenstern S, Strenov Y, Feinmesser M, Kravtsov V, Leon ME, Hajduch M, Ali SZ, VandenBussche CJ, Zhang X, Leider-Trejo L, Zubkov A, Vorobyov S, Kushnir M, Goren Y, Tabak S, Kadosh E, Benjamin H, Schnitzer-Perlman T, Marmor H, Motin M, Lebanony D, Kredo-Russo S, Mitchell H, Noller M, Smith A, Dattner O, Ashkenazi K, Sanden M, Berlin KA, Bar D, Meiri E. Multicentre validation of a microRNA-based assay for diagnosing indeterminate thyroid nodules utilising fine needle aspirate smears. J Clin Pathol. 2017 Jun;70(6):500-507. doi: 10.1136/jclinpath-2016-204089. Epub 2016 Oct 26. PMID 27798083